CLINICAL TRIAL: NCT06848127
Title: At the Frontier of Post-Traumatic Stress Disorder and Borderline Personality Disorder: Characterization Complex Post-traumatic Stress Disorder Via an Ecological, Physiological and Cognitive Approach to the Emotional Dysregulation
Brief Title: Study of Emotional Dysregulation in Complex Post-Traumatic Stress Disorder
Acronym: TR-EMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9362; 2024-A01240-47 (Other: ANSM)
Record Dates: First submitted 2025-02-12; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Complex Post-Traumatic Stress Disorder (CPTSD); Borderline Personality Disorder (BPD); Post-traumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Borderline Personality Disorder; Stress Disorders, Post-Traumatic | interventions — Mental Status and Dementia Tests; Ecological Momentary Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Healthy voluntary group (Active Comparator): 50 healthy volunteers who have been exposed to a traumatic event but without traumatic symptoms and with subthreshold scores on the PTSD Checklist for DSM-5 and Borderline Symptom List.
  Interventions: Other: Self-questionnaires; Other: Cognitive assessment; Other: Momentary Ecological Assessment (EMA)
- Group Patients with cPTSD (Experimental): 30 Patients diagnosed with cPTSD according to ICD-11 criteria
  Interventions: Other: Self-questionnaires; Other: Cognitive assessment; Other: Momentary Ecological Assessment (EMA); Other: Semi-structured interviews ITI and DSCID-II
- Group Patients with PTSD (Experimental): 30 Patients diagnosed with PTSD according to ICD-11 criteria
  Interventions: Other: Self-questionnaires; Other: Cognitive assessment; Other: Momentary Ecological Assessment (EMA); Other: Semi-structured interviews ITI and DSCID-II
- Group Patients with BPD (Experimental): 30 Patients with a diagnosis of BPD, according to DSM-5 criteria
  Interventions: Other: Self-questionnaires; Other: Cognitive assessment; Other: Momentary Ecological Assessment (EMA); Other: Semi-structured interviews ITI and DSCID-II
- Group Patients with cPTSD + BPD comorbidity (Experimental): 30 Patients with cPTSD + BPD comorbidity, established prior to inclusion
  Interventions: Other: Self-questionnaires; Other: Cognitive assessment; Other: Momentary Ecological Assessment (EMA); Other: Semi-structured interviews ITI and DSCID-II

INTERVENTIONS:
Other: Self-questionnaires — All subjects (healthy volunteers and all patients) will complete a battery of self-questionnaires, assessing emotional dysregulation, traumatic symptoms, alteration of the sense of self, sensitivity to social rejection, dissociative symptoms, child abuse, functional repercussions of the disorders, depressive and anxiety symptoms and Impulsivity.
Other: Cognitive assessment — Completion of cognitive assessment, consisting of verbal fluency tasks , emotional Hayling, a dissociative associative memory retrieval task, a negative priming task and a heart rhythm detection task. The tasks of associative-dissociative memory retrieval, negative priming and heart rhythm detection will be coupled with a physiological recording, via a Biopac, to measure the change in skin conductance, body temperature and heart rate. The negative priming task will also be associated with the recording of eye movements allowing an indirect measurement of attentional orientation.
Other: Momentary Ecological Assessment (EMA) — A momentary ecological evaluation protocol will be proposed (between visits V1 and V2 for all subjects and between V3 and V4 for the 4 groups of patients) in order to assess emotional and symptomatic dynamics in a daily life context through a connected wath. During 7 days, subjects will be invited, via their smartphone, to carry out daily semi-random readings (indicated by smartphone notifications) of their subjective emotional experiences (10 once/day), but also spontaneous (by reporting emotions deemed intense immediately afterwards that they take place).
Other: Semi-structured interviews ITI and DSCID-II — ITI International Trauma Interview is a semi-structured interview consisting of one part allocated to the description of a traumatic event and two parts addressing the symptoms of PTSD (i.e. reliving, avoidance and alteration of wakefulness) and the symptoms of the disturbance of self-organization.
  The SCID-II Structured Clinical Interview for DSM-IV Personality Disorder is a 90-item semi-structured interview, covering all 10 categories of personality disorder as described in the DSM-IV.
  Arms: Group Patients with BPD; Group Patients with PTSD; Group Patients with cPTSD; Group Patients with cPTSD + BPD comorbidity

SUMMARY:
This study aims to characterize emotional dysregulation in complex post-traumatic stress disorder (cPTSD) and to determine the extent to which it can promote the distinction with borderline personality disorder (BPD) and post-traumatic stress disorder (PTSD).

As emotional dysregulation is a dynamic process whose phenomenological manifestations are labile, associated with physiological modifications and modulated by cognitive processing, a multiple methodology associating measurements in a real-life ecological context with measurements performed in the hospital will be preferred.

Overall, this study proposes to capture, for the first time, the clinical manifestations associated with cPTSD from the perspective of emotional dysregulation and its underlying processes

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria common to healthy patients and volunteers: Subject, male or female, over 18 years of age; Subject able to understand the objectives and risks of the research and to give informed, dated and signed consent; Subject affiliated to a social protection health insurance scheme, beneficiary or beneficiary.
* Patient-specific inclusion criteria: Patient with a diagnosis of PTSD or PTSD according to ICD-11 criteria (World Health Organization, 2018). OR Patient with a diagnosis of BPD, according to DSM-5 criteria (American Psychiatric Association, 2013). OR Patient with cPTSD + BPD comorbidity, established prior to inclusion.
* Inclusion criteria specific to healthy volunteers: Subject who has been exposed to a traumatic event (Life Events Checklist, Gray et al., 2004) but without traumatic symptoms, or has subcut-off scores on PTSD scales (PCL-5, PTSD Checklist for DSM-5, Blevins et al., 2015), and TPB (BSL-23, Borderline Symptom List, Nicastro et al., 2016).

Exclusion Criteria:

* Non-inclusion criteria common to healthy patients and volunteers:

Subject who does not have a smartphone with an internet connection; Subject in an exclusion period (determined by a previous or ongoing study); Participation in another clinical study that may interfere with the study; Inability to provide the subject with informed information (subject in an emergency or life-threatening situation); Subject under the protection of justice; Subject under guardianship or curatorship; Pregnancy and/or breastfeeding.

-Patient-specific non-inclusion criteria: Patient with a diagnosis of a psychotic disorder (according to DSM-5 criteria, American Psychiatric Association, 2013); Patient with a diagnosis of severe substance use disorder (according to DSM-5 criteria, American Psychiatric Association, 2013); Patient with an intellectual disability (IQ ≤ 70); Patient with neurological (acquired brain injury) or neurovegetative comorbidity; Patient following or having undergone psychotherapy of the Dialectical Behavior Therapy (DBT) type; Patient with severe cardiac disorders; Patient on therapy that alters physiological response (e.g., beta-blockers).

-Specific non-inclusion criteria for healthy volunteers: Subject with a history of psychiatric, neurodevelopmental, neurological, neurovegetative or cardiac disorders; Subject on psychotropic therapy or treatment modifying physiological parameters (e.g., beta-blockers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Characterizing the emotional pattern | Day 1
  Comparison of DERS scores in groups ( an effect size of 0.37 for the means of DERS by group)

SECONDARY OUTCOMES:
Assessing subjective differences in real-life emotional experience | From Day 14 till Day 21
  Frequency of emotional responses observed in a real-life context. The subjective differences in real-life emotional experience between PTSD, PTSD, BPD, cPTSD + BPD and healthy volunteers, without traumatic symptoms, will be apprehended by an ecological momentary assessment protocol (EMA) . For 7 days, subjects will receive 10 daily notifications allowing them to inform their emotional experiences (m-Path application). The topics will complete a series of questions about emotions that have arisen since the last solicitation.
Evaluate physiological responses in hospital consultations and in real life | From Day 7 to Day 14
  Physiological parameters of emotion (skin conductance, body temperature and rhythm cardiac) between cPTSD, PTSD, BPD, PTSD+BPD and healthy volunteers, without traumatic symptoms, will be assessed from recording of different physiological parameters of emotion (heart rate, body temperature, skin conductance) made possible by the continuous wearing of a connected watch Empatica (EmbracePlus model, https://www.empatica.com/en-eu/embraceplus/) for 7 days. The physiological recording will be coupled with the subjective momentary ecological assessment.
Studying the cognitive correlates of emotional dysregulation | From Day 7 to Day 14
  Cognitive correlates of emotional dysregulation in CPTSD, PTSD, BPD, comorbid presentation of cPTSD + BPD and in healthy volunteers without traumatic symptoms will be assessed on the basis of several specific cognitive tests proposed during the visit of follow-up n°1 (V1).
Investigate the concordance between subjective and physiological measures of dysregulation Emotional | Up to 3 years
  The concordance between subjective, physiological and cognitive measures of dysregulation emotional studies collected in a real-life context (between V1 and V2) in patients (i.e. cPTSD, PTSD, BPD, cPTSD + BPD) and healthy volunteers, will be assessed from the correlation coefficients between frequency, intensity and emotional variability, conductance parameters body temperature and heart rate and response times and number of error to the emotional Stroop
The concordance between cognitive and physiological measures of dysregulation Emotional | Up to 3 years
  Coefficients of correlations between cognitive performance and physiological parameters. The concordance between cognitive and physiological measures, obtained in consultation, in patients (i.e. cPTSD, PTSD, BPD, cPTSD + BPD) and healthy volunteers, will be assessed from analyses correlations between performance (response times and errors) on each cognitive test and various physiological parameters recorded by the Biopac (carried out during a V1 visit).
The association between subjective and cognitive measures of emotional dysregulation | Up to 3 years
  Coefficients of correlations between self-questionnaire scores and performance Cognitive. The combination of subjective (self-questionnaires) and cognitive measures of dysregulation in patients (i.e. cPTSD, PTSD, BPD, cPTSD+BPD) and healthy volunteers, will be assessed on the basis of the correlation coefficients between the scores on the DERS, BEDS, PAQ and FREE and performance (response times and errors) at each cognitive test (fluences verbal, emotional hayling, negative priming task, memory recovery task associative-dissociative and heart rhythm detection task) carried out in visit V1).
Understand the entire clinical picture of cPTSD | Up to 3 years
  Scores obtained by subjects on supplementary questionnaires (i.e. not on emotional experience). The symptomatic characteristics of the different groups of subjects will be evaluated from their scores on the additional self questionnaires, proposed during the inclusion visit.
The evolution of self-reported emotional dysregulation after psychotherapeutic treatment in routine care | Up to 3 years
  Pre/Post Therapy Comparison of Dysregulation Self-Questionnaire Scores Emotional Following psychotherapy in routine care, it is expected that self-questionnaire scores on emotional dysregulation, namely DERS have significantly decreased in patients with cPTSD, PTSD, BPD, or cPTSD+BPD and significantly increased on the FREE scale. The investigators postulate that post-therapy scores of patients will be comparable to the scores of healthy subjects.
The evolution of emotional dynamics, assessed in daily life, after treatment psychotherapy in routine care | Up to 3 years
  Pre/Post Therapy Comparison of Frequency of Experiences emotional problems recorded in a real-life protocol (momentary ecological assessment, EMA).
The evolution of physiological emotional responses, assessed in daily life and in consultation, after psychotherapeutic treatment in routine care | Up to 3 years
  Pre/Post Therapy Comparison of the Physiological Parameters of Emotion Recorded by the Empatica EmbracePlus smartwatch.
Assessing subjective differences in real-life emotional experience | From Day 14 till Day 21
  Intensity and variability of emotional responses observed in a real-life context. The subjective differences in real-life emotional experience between PTSD, PTSD, BPD, cPTSD + BPD and healthy volunteers, without traumatic symptoms, will be apprehended by an ecological momentary assessment protocol (EMA). For 7 days, subjects will receive 10 daily notifications allowing them to inform their emotional experiences (m-Path application). The topics will complete a series of questions about emotions that have arisen since the last solicitation.
Assessing subjective differences in real-life emotional experience | From Day 14 till Day 21
  Variability of emotional responses observed in a real-life context. The subjective differences in real-life emotional experience between PTSD, PTSD, BPD, cPTSD + BPD and healthy volunteers, without traumatic symptoms, will be apprehended by an ecological momentary assessment protocol (EMA). For 7 days, subjects will receive 10 daily notifications allowing them to inform their emotional experiences (m-Path application). The topics will complete a series of questions about emotions that have arisen since the last solicitation.
Evaluate emotional responses in hospital consultations and in real life | From Day 7 to Day 14
  Physiological differences in emotional experiences between cPTSD, PTSD, BPD, PTSD+BPD and healthy volunteers, without traumatic symptoms, will be assessed from recording of the physiological parameters of the emotion will be made during the V1 visit to the University Hospitals of Strasbourg, in parallel with the taking of the tests via the Biopac wireless measurement system.
The evolution of self-reported emotional dysregulation after psychotherapeutic treatment in routine care | Up to 3 years
  Pre/Post Therapy Comparison of Dysregulation Self-Questionnaire Scores Emotional Following psychotherapy in routine care, it is expected that self-questionnaire scores on emotional dysregulation, namely BEDS have significantly decreased in patients with cPTSD, PTSD, BPD, or cPTSD+BPD and significantly increased on the FREE scale. The investigators postulate that post-therapy scores of patients will be comparable to the scores of healthy subjects.
The evolution of self-reported emotional dysregulation after psychotherapeutic treatment in routine care | Up to 3 years
  Pre/Post Therapy Comparison of Dysregulation Self-Questionnaire Scores Emotional Following psychotherapy in routine care, it is expected that self-questionnaire scores on emotional dysregulation, namely PAQ have significantly decreased in patients with cPTSD, PTSD, BPD, or cPTSD+BPD and significantly increased on the FREE scale. The investigators postulate that post-therapy scores of patients will be comparable to the scores of healthy subjects.
The evolution of emotional dynamics, assessed in daily life, after treatment psychotherapy in routine care | Up to 3 years
  Pre/Post Therapy Comparison of Intensity of Experiences emotional problems recorded in a real-life protocol (momentary ecological assessment, EMA).
The evolution of emotional dynamics, assessed in daily life, after treatment psychotherapy in routine care | Up to 3 years
  Pre/Post Therapy Comparison of Variability of Experiences emotional problems recorded in a real-life protocol (momentary ecological assessment, EMA).
The evolution of cognitive functioning underlying emotional dysregulation, after Psychotherapeutic treatment in routine care | Up to 3 years
  Pre/Post Therapy Comparison of Performance in Verbal Fluency Tests emotional and autobiographical, to the emotional Hayling.
The evolution of cognitive functioning underlying emotional dysregulation, after Psychotherapeutic treatment in routine care | Up to 3 years
  Pre/Post Therapy Comparison of Performance in Verbal Fluency Tests emotional and autobiographical, to a negative priming task.
The evolution of cognitive functioning underlying emotional dysregulation, after Psychotherapeutic treatment in routine care | Up to 3 years
  Pre/Post Therapy Comparison of Performance in Verbal Fluency Tests emotional and autobiographical to the Heart Rhythm Detection Task.
The evolution of cognitive functioning underlying emotional dysregulation, after Psychotherapeutic treatment in routine care | Up to 3 years
  Pre/Post Therapy Comparison of Performance in Verbal Fluency Tests emotional and autobiographical to an Emotional Stroop.

CONTACTS AND LOCATIONS:
Overall Officials: Luisa WEINER, Professor, Principal Investigator — Department of Psychiatry II Psychiatry, Mental Health and Addiction Medicine, University Hospitals of Strasbourg